CLINICAL TRIAL: NCT05779514
Title: Effect of Mirabegron on Promoting Brown Adipose Tissue Activation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zhejiang Provincial People's Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: YJKY20220007
Record Dates: First submitted 2023-02-16; First posted 2023-03-22 (Actual); Last update posted 2023-03-22 (Actual); Status verified 2023-03

CONDITIONS: Tumour
Keywords: brown adipose tissue; Mirabegron
MeSH Terms: conditions — Neoplasms | interventions — mirabegron

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- The growth of brown adipose tissue (Experimental)
  Interventions: Drug: Mirabegron

INTERVENTIONS:
Drug: Mirabegron — Health Volunteers ：Mirabegron p.o. 28 days 100mg qd./ Tumor patients ：Mirabegron p.o. 28 days 100 mg qd or 200 mg qd.

SUMMARY:
In previous preclinical studies, our group found that Mirabegron, a clinical drug, could activate brown adipose tissue and inhibit tumor growth in tumour-bearing mice.Investigators look forward to further evaluating the effect of Mirabegron-mediated brown adipose tissue activation, so as to provide new drug applications for clinical cancer prevention and treatment

ELIGIBILITY:
Inclusion Criteria:

* Health Volunteers

  1. Sign the informed consent before the study, and fully understand the content, process and possible adverse events.
  2. Both men and women, aged 18-75 years (including the boundary value) .
  3. Body mass index (BMI) is 19.0-26.0 kg/m2 (including the boundary value).
* Tumor patients

  1. Sign the informed consent before the study, and fully understand the content, process and possible adverse events.
  2. Tumor bearing and not in the period of chemotherapy and targeted drug intervention).
  3. Both men and women, aged 18-75 years (including the boundary value) .
  4. Body mass index (BMI) is 19.0-26.0 kg/m2 (including the boundary value).
  5. Proper bone marrow and organ function, as defined below:HB≥80h/L; ANC≥1.5*109/L; PLT≥50*109/L; ALT≤3 upper limit of normal ( ULN ); AST≤3 ULN ; TBIL≤1.5 ULN.
  6. The expected survival is 3 months or more.

Exclusion Criteria:

* Health Volunteers and Tumor patients

  1. A history of tuberculosis infection.
  2. Patients with contraindications to Mirabegron: allergic to Mirabegron or any of its excipients; Patients with poorly controlled severe hypertension(SBP≧180mmHg or/and DBP≧110mmHg).
  3. Women who are pregnant or breastfeeding.
  4. The subject may not be able to complete the study for other reasons or may not be able to participate in the study for other reasons judged by the investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2022-08-18 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
The growth of brown adipose tissue by PET-CT | Day 0 and Day 28
  Growth of brown adipose tissue after 28 days of oral administration of Mirabegron was measured by standard uptake value (SUV) values measured by PET-CT .

SECONDARY OUTCOMES:
blood glucose and glucose tolerance test ( GTT ) by Hematological tests | Day 0 and Day 28
  The change of glucose( mmol/L ) and glucose tolerance test( mmol/L ) after 28 days of oral administration of Mirabegron by Hematological tests .

CONTACTS AND LOCATIONS:
Overall Officials: Minghua Ge, Doctor, Study Chair — Institution Affiliation
Locations (1):
- Zhejiang Provincial People's Hospital, Hangzhou, Zhejiang, China